CLINICAL TRIAL: NCT05730725
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Phase 2 Study to Evaluate the Clinical Efficacy and Safety of BMS-986322 in Participants With Moderate-to-Severe Psoriasis
Brief Title: A Study to Evaluate Effectiveness and Safety of BMS-986322 in Participants With Moderate-to-Severe Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM032-041; 2023-504848-34 (EudraCT Number); U1111-1282-3606 (Registry Identifier: WHO)
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Results first posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Psoriasis
Keywords: Moderate-to-Severe Psoriasis; BMS-986322; TYK2 inhibitor
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BMS-986322 Dose 1 (Experimental)
  Interventions: Drug: BMS-986322
- BMS-986322 Dose 2 (Experimental)
  Interventions: Drug: BMS-986322
- BMS-986322 Dose 3 (Experimental)
  Interventions: Drug: BMS-986322
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BMS-986322 — Specified dose on specified days
  Arms: BMS-986322 Dose 1; BMS-986322 Dose 2; BMS-986322 Dose 3
Other: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate clinical effectiveness and safety of BMS-986322 in participants with moderate-to-severe psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of plaque psoriasis (PsO) for ≥ 6 months
* Body mass index 18 to 40 kg/m^2 and total body weight > 50 kg (110 lbs)
* Deemed by Investigator to be eligible for phototherapy or systemic therapy
* Psoriatic plaques must cover ≥ 10% of body surface area at baseline
* Psoriasis Area and Severity Index (PASI) score ≥ 12 and static Physician Global Assessment (sPGA) ≥ 3 at baseline

Exclusion Criteria:

* Diagnosis of non-plaque psoriasis (guttate, inverse, pustular, erythrodermic)
* Diagnosis of uveitis, inflammatory bowel disease, or other immune-mediated conditions that are commonly associated with PsO for which a participant requires current systemic immunosuppressant medical treatment
* Any significant acute or chronic medical illness

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (35):
- United States (19):
  - Local Institution - 0006, Birmingham, Alabama
  - Local Institution - 0012, Encino, California
  - Local Institution - 0005, Fountain Valley, California
  - Local Institution - 0002, Fremont, California
  - Local Institution - 0001, Los Angeles, California
  - Local Institution - 0016, Los Angeles, California
  - Local Institution - 0003, Santa Ana, California
  - Local Institution - 0013, Coral Gables, Florida
  - Local Institution - 0056, Skokie, Illinois
  - Local Institution - 0044, Clarksville, Indiana
  - Local Institution - 0057, Leawood, Kansas
  - Local Institution - 0004, Beverly, Massachusetts
  - Local Institution - 0060, Lee's Summit, Missouri
  - Local Institution - 0007, Portsmouth, New Hampshire
  - Local Institution - 0055, Durham, North Carolina
  - Local Institution - 0008, Cleveland, Ohio
  - Local Institution - 0058, Rapid City, South Dakota
  - Local Institution - 0059, Dallas, Texas
  - Local Institution - 0011, Webster, Texas
- Australia (3):
  - Local Institution - 0024, Brisbane, Queensland
  - Local Institution - 0019, Carlton, Victoria
  - Local Institution - 0045, Pascoe Vale South, Victoria
- Canada (5):
  - Local Institution - 0062, St. John's, Newfoundland and Labrador
  - Local Institution - 0034, Barrie, Ontario
  - Local Institution - 0020, Hamilton, Ontario
  - Local Institution - 0041, London, Ontario
  - Local Institution - 0030, Toronto, Ontario
- Japan (6):
  - Local Institution - 0049, Sapporo, Hokkaido
  - Local Institution - 0023, tabashi City, Tokyo
  - Local Institution - 0051, Fukuoka
  - Local Institution - 0042, Itabashi-Ku
  - Local Institution - 0026, Nagoya
  - Local Institution - 0027, Tsu
- United Kingdom (2):
  - Local Institution - 0050, Hinckley, LEC
  - Local Institution - 0046, Leytonstone

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trialsand research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 109 Participants Enrolled and Treated
Groups:
- Placebo: Placebo
- Treatment 1: BMS-986322 16mg
- Treatment 2: BMS-986322 32mg
- Treatment 3: BMS-986322 64mg
Period: Overall Study
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3
Started | 28 | 27 | 27 | 27
Completed | 24 | 26 | 26 | 25
Not Completed | 4 | 1 | 1 | 2
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 1
Not completed — Not Reported | 1 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3 | Total
Number analyzed (Participants) | 28 | 27 | 27 | 27 | 109
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.1 (10.77) | 50.2 (14.31) | 50.8 (10.82) | 45.9 (12.09) | 49.5 (12.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 9 | 7 | 35
  Male | 20 | 16 | 18 | 20 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 12 | 8 | 8 | 39
  Not Hispanic or Latino | 16 | 15 | 18 | 19 | 68
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 1 | 2 | 6
  Asian | 7 | 7 | 4 | 6 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 3 | 5
  White | 18 | 18 | 21 | 16 | 73
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achiving PASI-75 at Week 12
Description: PASI is a measure of the average erythema, induration thickness, and scaling of psoriatic skin lesions (each graded on a 0 to 4 scale), weighted by the area of involvement (head, arms, trunk to groin, and legs to top of buttocks).
  The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity.
  The PASI-75 response rate is defined as the percentage of participants with moderate-to-severe PsO achieving at least 75% reduction from baseline in PASI score.
  Baseline is defined as the last measurement on or prior to date/time of first dose of study treatment.
Time Frame: 12 Weeks
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3
Number analyzed (Participants) | 28 | 23 | 26 | 27
Percentage | 3.6 [0.1 to 18.3] | 47.8 [26.8 to 69.4] | 80.8 [60.6 to 93.4] | 63.0 [42.4 to 80.6]

2. Primary Outcome: Number of Participants With Safety Related Events
Description: Treatment related adverse events, serious adverse events and treatment related adverse events leading to treatment discontinuation are considered safety related events.
Time Frame: approximately 85 days
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3
Number analyzed (Participants) | 28 | 27 | 27 | 27
Participants
  Any TEAE | 16 | 14 | 14 | 16
  Any SAE | 1 | 1 | 0 | 0
  TEAEs leading to discontinuation | 2 | 0 | 0 | 1

3. Primary Outcome: Number of Participants With TEAE by Worst Intensity
Description: Mild TEAE: An event that is easily tolerated by the participant, causing minimal discomfort, and not interfering with everyday activities.
  Moderate TEAE:An event that causes sufficient discomfort and interferes with normal everyday activities.
  Severe TEAE: An event that prevents normal everyday activities. An AE that is assessed as severe should not be confused with an SAE. Severe is a category utilized for rating the intensity of an event, and both AEs and SAEs can be assessed as severe.
Time Frame: approximately 5 months
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3
Number analyzed (Participants) | 28 | 27 | 27 | 27
Participants
  Mild | 10 | 7 | 10 | 10
  Moderate | 6 | 7 | 4 | 6
  Severe | 0 | 0 | 0 | 0
  Not Reported | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With AE Indicating Clinical Laboratory Abnormality
Description: Number of participants with AE indicating clinical laboratory abnormality
Time Frame: approximately 5 months
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3
Number analyzed (Participants) | 28 | 27 | 27 | 27
Participants
  Hypercholesterolaemia | 0 | 0 | 1 | 0
  Hypernatraemia | 0 | 0 | 0 | 1
  Anaemia | 0 | 0 | 0 | 1
  Iron Deficiency Anaemia | 0 | 0 | 0 | 1
  Thrombocytopenia | 0 | 0 | 0 | 1
  Hyertransaminasaemia | 0 | 0 | 0 | 1
  Blood creatine phosphokinase increased | 0 | 1 | 0 | 0

5. Secondary Outcome: Percentage of Participants Achiving sPGA Score of 0 or 1 at Week 12
Description: The static Physician's Global Assessment(sPGA)
  The sPGA is used to assess a participant's psoriasis lesions at a specific time point. Lesions are graded based on three characteristics:
  Erythema (E) Induration (I) Scaling (S)
  Each is scored individually, and the average of the three scores, rounded to the nearest whole number, determines the final sPGA score.
  0 = No evidence
  1= Minimal 2 = Mild 3 = Moderate 4 = Severe.
  The lower the score the better.
Time Frame: 12 Weeks
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3
Number analyzed (Participants) | 28 | 24 | 26 | 27
Percentage | 3.6 [0.1 to 18.3] | 54.2 [2.8 to 74.4] | 69.2 [48.2 to 85.7] | 55.6 [35.3 to 74.5]

6. Secondary Outcome: Percentage of Participants Achiving PASI-50 at Week 12
Description: PASI is a measure of the average erythema, induration thickness, and scaling of psoriatic skin lesions (each graded on a 0 to 4 scale), weighted by the area of involvement (head, arms, trunk to groin, and legs to top of buttocks).
  The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity.
  The PASI-50 response rate is defined as the percentage of participants with moderate-to-severe PsO achieving at least 50% reduction from baseline in PASI score.
  Baseline is defined as the last measurement on or prior to date/time of first dose of study treatment.
Time Frame: 12 Weeks
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3
Number analyzed (Participants) | 28 | 23 | 26 | 27
Percentage of Participants | 17.9 [6.1 to 36.9] | 73.9 [51.6 to 89.8] | 92.3 [74.9 to 99.1] | 81.5 [61.9 to 93.7]

7. Secondary Outcome: Percentage of Participants Achiving PASI-90 at Week 12
Description: PASI is a measure of the average erythema, induration thickness, and scaling of psoriatic skin lesions (each graded on a 0 to 4 scale), weighted by the area of involvement (head, arms, trunk to groin, and legs to top of buttocks).
  The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity.
  The PASI-90 response rate is defined as the percentage of participants with moderate-to-severe PsO achieving at least 90% reduction from baseline in PASI score.
  Baseline is defined as the last measurement on or prior to date/time of first dose of study treatment.
Time Frame: 12 Weeks
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3
Number analyzed (Participants) | 28 | 23 | 26 | 27
Percentage of Participants | 3.6 [0.1 to 18.3] | 13.0 [2.8 to 33.6] | 61.5 [40.6 to 79.8] | 40.7 [22.4 to 61.2]

8. Secondary Outcome: Percentage of Participants Achiving PASI-100 at Week 12
Description: PASI is a measure of the average erythema, induration thickness, and scaling of psoriatic skin lesions (each graded on a 0 to 4 scale), weighted by the area of involvement (head, arms, trunk to groin, and legs to top of buttocks).
  The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity.
  The PASI-100 response rate is defined as the percentage of participants with moderate-to-severe PsO achieving at least 100% reduction from baseline in PASI score.
  Baseline is defined as the last measurement on or prior to date/time of first dose of study treatment.
Time Frame: 12 Weeks
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3
Number analyzed (Participants) | 28 | 23 | 26 | 27
Percentage of Participants | 0 [0.0 to 12.3] | 0 [0.0 to 14.8] | 15.4 [4.4 to 34.9] | 3.7 [0.1 to 19.0]

9. Secondary Outcome: Change of PASI-75 Scores Overtime
Description: as for outcome 1
Time Frame: From start of treatment (Week 1) to Week 2, 4, 8 and 12
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3
Number analyzed (Participants) | 28 | 27 | 27 | 27
Percentage of Participants
  Week 1: number analyzed (Participants) | 25 | 26 | 26 | 26
  Week 1 | 0.0 [0.0 to 13.7] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 13.2] | 3.8 [0.1 to 19.6]
  Week 2: number analyzed (Participants) | 25 | 27 | 26 | 25
  Week 2 | 0.0 [0.0 to 13.7] | 0.0 [0.0 to 12.8] | 11.5 [2.4 to 30.2] | 4.0 [0.1 to 20.4]
  Week 4: number analyzed (Participants) | 28 | 27 | 27 | 26
  Week 4 | 3.6 [0.1 to 18.3] | 7.4 [0.9 to 24.3] | 33.3 [16.5 to 54.0] | 30.8 [14.3 to 51.8]
  Week 8: number analyzed (Participants) | 25 | 25 | 27 | 26
  Week 8 | 4.0 [0.1 to 20.4] | 40.0 [21.1 to 61.3] | 66.7 [46.0 to 83.5] | 57.7 [36.9 to 76.6]
  Week 12: number analyzed (Participants) | 24 | 22 | 26 | 25
  Week 12 | 4.2 [0.1 to 21.1] | 54.5 [32.2 to 75.6] | 80.8 [60.6 to 93.4] | 72.0 [50.6 to 87.9]

10. Secondary Outcome: Change of PASI-90 Scores Overtime
Description: as for outcome 7
Time Frame: From start of treatment (Week 1) to Week 2, 4, 8 and 12
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3
Number analyzed (Participants) | 28 | 27 | 27 | 27
Percentage of Participants
  Week 1: number analyzed (Participants) | 25 | 26 | 26 | 26
  Week 1 | 0.0 [0.0 to 13.7] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 13.2]
  Week 2: number analyzed (Participants) | 25 | 27 | 26 | 25
  Week 2 | 0.0 [0.0 to 13.7] | 0.0 [0.0 to 12.8] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 13.7]
  Week 4: number analyzed (Participants) | 28 | 27 | 27 | 26
  Week 4 | 0.0 [0.0 to 12.3] | 0.0 [0.0 to 12.8] | 18.5 [6.3 to 38.1] | 7.7 [0.9 to 25.1]
  Week 8: number analyzed (Participants) | 25 | 25 | 27 | 26
  Week 8 | 4.0 [0.1 to 20.4] | 8.0 [1.0 to 26.0] | 25.9 [11.1 to 46.3] | 30.8 [14.3 to 51.8]
  Week 12: number analyzed (Participants) | 24 | 22 | 26 | 25
  Week 12 | 4.2 [0.1 to 21.1] | 13.6 [2.9 to 34.9] | 61.5 [40.6 to 79.8] | 48.0 [27.8 to 68.7]

11. Secondary Outcome: Change of PASI-100 Scores Overtime
Description: as for outcome 8
Time Frame: From start of treatment (Week 1) to Week 2, 4, 8 and 12
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3
Number analyzed (Participants) | 28 | 27 | 27 | 27
Percentage of Participants
  Week 1: number analyzed (Participants) | 25 | 26 | 26 | 26
  Week 1 | 0.0 [0.0 to 13.7] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 13.2]
  Week 2: number analyzed (Participants) | 25 | 27 | 26 | 25
  Week 2 | 0.0 [0.0 to 13.7] | 0.0 [0.0 to 12.8] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 13.7]
  Week 4: number analyzed (Participants) | 28 | 27 | 27 | 26
  Week 4 | 0.0 [0.0 to 12.3] | 0.0 [0.0 to 12.8] | 3.7 [0.1 to 19.0] | 0.0 [0.0 to 13.2]
  Week 8: number analyzed (Participants) | 25 | 25 | 27 | 26
  Week 8 | 0.0 [0.0 to 13.7] | 0.0 [0.0 to 13.7] | 3.7 [0.1 to 19.0] | 0.0 [0.0 to 13.2]
  Week 12: number analyzed (Participants) | 24 | 22 | 26 | 25
  Week 12 | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 15.4] | 15.4 [4.4 to 34.9] | 4.0 [0.1 to 20.4]

12. Secondary Outcome: Change of PASI-50 Scores Overtime
Description: as for outcome 6
Time Frame: From start of treatment (Week 1) to Week 2, 4, 8 and 12
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3
Number analyzed (Participants) | 28 | 27 | 27 | 27
Percentage of Participants
  Week 1: number analyzed (Participants) | 25 | 26 | 26 | 26
  Week 1 | 0.0 [0.0 to 13.7] | 3.8 [0.1 to 19.6] | 7.7 [0.9 to 25.1] | 7.7 [0.9 to 25.1]
  Week 2: number analyzed (Participants) | 25 | 27 | 26 | 25
  Week 2 | 12.0 [2.5 to 31.2] | 14.8 [4.2 to 33.7] | 34.6 [17.2 to 55.7] | 24.0 [9.4 to 45.1]
  Week 4: number analyzed (Participants) | 28 | 27 | 27 | 26
  Week 4 | 10.7 [2.3 to 28.2] | 48.1 [28.7 to 68.1] | 66.7 [46.0 to 83.5] | 65.4 [44.3 to 82.8]
  Week 8: number analyzed (Participants) | 25 | 25 | 27 | 26
  Week 8 | 8.0 [1.0 to 26.0] | 84.0 [63.9 to 95.5] | 85.2 [66.3 to 95.8] | 88.5 [69.8 to 97.6]
  Week 12: number analyzed (Participants) | 24 | 22 | 26 | 25
  Week 12 | 20.8 [7.1 to 42.2] | 81.8 [59.7 to 94.8] | 92.3 [74.9 to 99.1] | 92.0 [74.0 to 99.0]

13. Secondary Outcome: Mean Change Frome Baseline of PASI Scores Overtime
Description: PASI is a measure of the average erythema, induration thickness, and scaling of psoriatic skin lesions (each graded on a 0 to 4 scale), weighted by the area of involvement (head, arms, trunk to groin, and legs to top of buttocks).
  The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity.
  Baseline is defined as the last measurement on or prior to date/time of first dose of study treatment.
Time Frame: From start of treatment (Week 1) to Week 2, 4, 8, and 12
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: PASI Score on a Scale
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3
Number analyzed (Participants) | 28 | 27 | 27 | 27
PASI Score on a Scale
  Week 1: number analyzed (Participants) | 25 | 26 | 26 | 26
  Week 1 | -0.50 (5.765) | -2.85 (3.782) | -2.95 (4.525) | -3.36 (4.047)
  Week 2: number analyzed (Participants) | 25 | 27 | 26 | 25
  Week 2 | -3.30 (5.803) | -5.16 (4.856) | -7.13 (6.699) | -6.27 (5.421)
  Week 4: number analyzed (Participants) | 28 | 27 | 27 | 26
  Week 4 | -3.97 (7.872) | -8.53 (6.311) | -10.63 (7.512) | -10.05 (6.629)
  Week 8: number analyzed (Participants) | 25 | 25 | 27 | 26
  Week 8 | -3.73 (7.521) | -13.34 (5.734) | -13.66 (8.265) | -14.06 (6.452)
  Week 12: number analyzed (Participants) | 24 | 22 | 26 | 25
  Week 12 | -4.43 (8.030) | -14.55 (6.644) | -15.39 (8.971) | -15.44 (6.429)

14. Secondary Outcome: Ctrough Measurements Overtime
Description: trough observed plasma concentration
Time Frame: From start of treatment (Week 1) to Week 2, 4, 8 and 12
Population: All participants who were treated with BMS-986322 and with PK measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3
Number analyzed (Participants) | 27 | 27 | 27
ng/mL
  Week 1: number analyzed (Participants) | 25 | 21 | 20
  Week 1 | 55.463 (83.8) | 128.971 (121.6) | 138.950 (735.3)
  Week 2: number analyzed (Participants) | 24 | 20 | 19
  Week 2 | 57.595 (97.7) | 99.871 (273.3) | 191.509 (349.3)
  Week 4: number analyzed (Participants) | 23 | 20 | 22
  Week 4 | 57.728 (73.7) | 111.379 (235.3) | 153.285 (618.6)
  Week 8: number analyzed (Participants) | 20 | 21 | 23
  Week 8 | 42.370 (224.9) | 68.035 (479.9) | 112.852 (1125.2)
  Week 12: number analyzed (Participants) | 20 | 22 | 20
  Week 12 | 47.321 (235.6) | 52.295 (534.0) | 82.047 (3201.7)

15. Secondary Outcome: Cmax at Day 15
Description: maximum observed concentration
Time Frame: At Day 15 post first dose
Population: All participants who were treated with BMS-986322 and with Cmax measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3
Number analyzed (Participants) | 25 | 24 | 23
ng/mL | 210.410 (36.1) | 411.027 (41.9) | 871.064 (34.9)

16. Secondary Outcome: Tmax at Day 15
Description: time to maximum observed concentration
Time Frame: At Day 15 post first dose
Population: All participants who were treated with BMS-986322 and with Tmax measurements
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3
Number analyzed (Participants) | 25 | 24 | 23
hours | 1.0830 [0.500 to 5.000] | 1.0415 [0.000 to 5.050] | 2.000 [0.917 to 4.750]

17. Secondary Outcome: AUC(Tau) at Day 15
Description: area under the plasma concentration-time curve over the dosing interval
Time Frame: At Day 15 post first dose
Population: All participants who were treated with BMS-986322 and with AUC(Tau) measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3
Number analyzed (Participants) | 25 | 24 | 22
h*ng/mL | 2576.824 (49.3) | 5057.790 (53.2) | 11815.731 (37.1)

18. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in ECG Evaluations.
Description: Number of participants with clinically significant changes from baseline in ECG evaluations.
  ECG results for participants with any result outside of a pre-specified range and investigator identified abnormalities will be listed for the Safety Population.
  The following criteria will be used to determine ECG results that are outside of a pre-specified range:
  * PR (msec): Value > 200
  * QRS (msec): Value > 120
  * QT (msec): Value > 500 or change from baseline > 30
  * QTcF (msec): Value > 450 or change from baseline > 30
Time Frame: approximately 5 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3
Number analyzed (Participants) | 28 | 27 | 27 | 27
Participants | 0 | 0 | 0 | 0

19. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Vital Signs Evaluations
Description: Number of participants with clinically significant changes from baseline in vital signs evaluations.
  Vital signs for participants with any out-of-range result will be listed for the Safety Population.
  The following criteria will be used to determine vital sign results that are outside of a prespecified range, where changes from baseline are based on matched postural positions:
  * Heart Rate (bpm): Value > 100 and change from baseline > 30, or Value < 55 and change from baseline < -15
  * Systolic blood pressure (mmHg): Value > 140 and change from baseline > 20, or Value < 90 and change from baseline < -20
  * Diastolic blood pressure (mmHg): Value > 90 and change from baseline > 10, or Value < 55 and change from baseline < -10
  * Respiration (breaths/min): Value > 16 or change from baseline > 10
  * Temperature (°C): Value > 38.3 or change from baseline > 1.6
Time Frame: approximately 5 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3
Number analyzed (Participants) | 28 | 27 | 27 | 27
Participants | 0 | 0 | 0 | 0

20. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Physical Examination Evaluations
Description: Number of participants with clinically significant changes from baseline in physical examination evaluations
Time Frame: approximately 5 months
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3
Number analyzed (Participants) | 28 | 27 | 27 | 27
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events, Serious Adverse Events:,All-Cause mortality (From randomization to end of study treatment): Approximately 85 Days
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Groups:
- Treatment 1: BMS-986322 16 mg
- Treatment 2: BMS-986322 32 mg
- Treatment 3: BMS-986322 64 mg
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/27 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/28 | 1/27 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 7/28 | 7/27 | 10/27 | 11/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=28) | Treatment 1 (N=27) | Treatment 2 (N=27) | Treatment 3 (N=27)
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=28) | Treatment 1 (N=27) | Treatment 2 (N=27) | Treatment 3 (N=27)
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 3
Folliculitis (Infections and infestations) | 0 | 0 | 3 | 0
Herpes zoster (Infections and infestations) | 2 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 2 | 1 | 2
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 2 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 4
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 4 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/25/NCT05730725/Prot_SAP_000.pdf